CLINICAL TRIAL: NCT01567605
Title: Bowel Care and Cardiovascular Function After Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Victoria Claydon, Assistant Professor, Simon Fraser University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011s0593
Record Dates: First submitted 2012-03-23; First posted 2012-03-30 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; autonomic dysreflexia; blood pressure; bowel care management; defecation
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine lubricant (then placebo) (Experimental): In this arm, on the first test day subjects will use lidocaine lubricant in their normal bowel care routine (rather than standard lubricating jelly). After a washout period they will repeat testing with the placebo lubricant.
  Interventions: Drug: Lidocaine lubricant; Other: Placebo lubricant
- Placebo lubricant (then lidocaine) (Placebo Comparator): In this arm, on the first test day subjects will use regular lubricant (AMG MedPro lubricating gel) in their normal bowel care routine. After a washout period they will repeat testing with a the lidocaine lubricant.
  Interventions: Drug: Lidocaine lubricant; Other: Placebo lubricant

INTERVENTIONS:
Drug: Lidocaine lubricant — Subjects using this intervention will receive 30 mL of Lidocaine hydrochloride jelly (2%)
  Other Names: xylocaine jelly (2%) AstraZeneca
Other: Placebo lubricant — Subjects using this intervention will receive 30 mL of placebo lubricant (no topical anesthetic)
  Other Names: AMG MedPro lubricating Gel

SUMMARY:
The main goal of this project is to determine the effects of lidocaine lubricant on cardiovascular function during routine bowel care in individuals with spinal cord injury. Bowel care is a common trigger of blood pressure and heart rate changes after spinal cord injury. In this project, we will be measuring blood pressure and heart rate non-invasively during normal bowel routine (which can be performed in the subject's home or at one of the investigators facilities). The measurements will occur twice over a period of 28 days: once using lidocaine lubricant and once using normal (placebo) lubricant. The recording equipment will be attached and subjects will have complete privacy during their bowel routine. The trial will be double-blind, meaning that neither the subject or the Nurse Continence Advisor who assists with testing will know which lubricant is being used for each test.

The use of a lubricant gel containing an anesthetic is the standard of care in many hospital facilities when performing bowel care for individuals with spinal cord injury; however, it is not often used in the home setting. It is thought that using anaesthetic might reduce the cardiovascular effects of bowel care after spinal cord injury. However, it is not known whether this is the case.

The investigators hypothesize that the lidocaine lubricant will alleviate some of the blood pressure and heart rate changes that occur during bowel care.

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate the effects of topical anesthesia on cardiovascular changes triggered by bowel care in people with spinal cord injury.

In people with spinal cord injury, episodes of high blood pressure are common during strong sensory stimuli such as those present during routine bowel care. These episodes of high blood pressure can be dangerous due to the magnitude of blood pressure increase and because they can be accompanied by irregular heart beats. This condition, known as autonomic dysreflexia, is most common in individuals with high-level injuries.

The experience of autonomic dysreflexia can vary widely between individuals: some have goosebumps, sweating, facial flushing or headaches, while others have no symptoms at all, despite their changes in heart rate and blood pressure.

The use of a lubricant gel containing an anesthetic, lidocaine lubricant, is the standard of care in many hospital facilities when performing bowel care for individuals with spinal cord injury; however, it is not often used in the home setting. It is thought that using anaesthetic might reduce the cardiovascular effects of bowel care after spinal cord injury. However, it is not known whether this is the case. We do not yet know the long-term consequences of these short-term elevations in blood pressure during autonomic dysreflexia, but given that they are often associated with discomfort, and have been known to be associated with more severe events such as stroke, it would be beneficial to reduce their occurrence.

Therefore, we will test whether lidocaine lubricant compared to a placebo lubricant improves the symptoms and signs of autonomic dysreflexia during bowel care in people with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* traumatic spinal cord injury at least one year ago
* regular bowel care routine (at least four weeks)

Exclusion Criteria:

* cauda equina or conus lesion
* currently use ventilator
* colostomy, or do not perform regular bowel care for any reason
* any skin breakdown (pressure sores)
* do not speak English
* are under 19 years old
* are pregnant or think you might be pregnant
* medical/psychiatric condition or substance abuse that is likely to affect your ability to complete this study
* currently using medications containing lidocaine
* allergy to lidocaine

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria E Claydon, PhD, Principal Investigator — Simon Fraser University and International Collaboration on Repair Discoveries (ICORD)
Locations (2):
- Canada (2):
  - Simon Fraser University, Burnaby, British Columbia
  - International Collaboration on Repair Discoveries, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (n=13) were recruited using a multi-method approach. Print advertisements were circulated through our community partner, Spinal Cord Injury British Columbia, via their quarterly publication, The Spin, and online advertisements were posted through our institutional website (www.icord.org).
Pre-assignment Details: All participants met eligibility criteria and were randomised to treatment in a crossover manner.
Groups:
- Lidocaine Lubricant (1 Day) Followed by Placebo Lubricant (1 Day): In this arm, subjects will first use lidocaine lubricant in their normal bowel care routine and then standard lubricant jelly.
  Lidocaine lubricant: Subjects using this intervention will receive 30 mL of Lidocaine hydrochloride jelly (2%) on test day one and 30mL of placebo lubricant jelly (AMG MedPro lubricating gel) on day two.
- Placebo Lubricant (1 Day) Followed by Lidocaine Lubricant (1 Day): In this arm, subjects will use placebo lubricant (AMG MedPro lubricating gel) in their normal bowel care routine on test day one followed by 30 mL of Lidocaine hydrochloride jelly (2%) on test day two.
Period: Overall Study
Arm/Group | Lidocaine Lubricant (1 Day) Followed by Placebo Lubricant (1 Day) | Placebo Lubricant (1 Day) Followed by Lidocaine Lubricant (1 Day)
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine Lubricant Then Placebo Lubricant: In this arm, subjects will use lidocaine lubricant in their normal bowel care routine on test day one and placebo lubricant on test day two.
  Lidocaine lubricant: Subjects using this intervention will receive 30 mL of Lidocaine hydrochloride jelly (2%).
  Placebo lubricant: Subjects using this intervention will receive 30 mL of placebo lubricant (no topical anesthetic)
- Placebo Lubricant Then Lidocaine Lubricant: In this arm, subjects will use placebo lubricant (AMG MedPro lubricating gel) in their normal bowel care routine on test day one and lidocaine lubricant on test day two.
  Placebo lubricant: Subjects using this intervention will receive 30 mL of placebo lubricant (no topical anesthetic)
  Lidocaine lubricant: Subjects using this intervention will receive 30 mL of Lidocaine hydrochloride jelly (2%)
- Total: Total of all reporting groups
Arm/Group | Lidocaine Lubricant Then Placebo Lubricant | Placebo Lubricant Then Lidocaine Lubricant | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11) | 47 (14) | 44 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Change During Bowel Care
Description: Beat-to-beat blood pressure will be recorded using a finger blood pressure cuff (Finometer) on two occasions within 28 days, for up to one hour on each occasion.
Time Frame: Measured continuously during bowel care (approximately one hour) on two occasions within 28 days.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Lidocaine Lubricant: In this arm, subjects will use lidocaine lubricant in their normal bowel care routine (rather than standard lubricating jelly).
  Lidocaine lubricant: Subjects using this intervention will receive 30 mL of Lidocaine hydrochloride jelly (2%)
- Placebo Lubricant: In this arm, subjects will use regular lubricant (AMG MedPro lubricating gel) in their normal bowel care routine.
  Placebo lubricant: Subjects using this intervention will receive 30 mL of placebo lubricant (no topical anesthetic)
Arm/Group | Lidocaine Lubricant | Placebo Lubricant
Number analyzed (Participants) | 13 | 13
mmHg | 90.5 (13.4) | 80 (8.7)

2. Secondary Outcome: Duration of Bowel Care Routine
Description: The duration of bowel care routine will be recorded on two occasions within 28 days.
Time Frame: The exact duration of bowel care will be noted on two days within a 28 day period
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Lidocaine Lubricant | Placebo Lubricant
Number analyzed (Participants) | 13 | 13
minutes | 79.1 (10) | 57.7 (6.3)

3. Secondary Outcome: Cardiovascular Symptoms During Bowel Care
Description: Cardiovascular symptoms will be recorded using a questionnaire on two occasions within 28 days. The questionnaire takes approximately 15 minutes to complete. The symptom score rated 13 measures (from 0-4) based on the frequency of symptoms experiences with a possible score ranging from 0-52. High scores denote more severe symtoms.
Time Frame: Measured by questionnaire (approximately 15 minutes) after bowel care on two occasions within 28 days.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lidocaine Lubricant | Placebo Lubricant
Number analyzed (Participants) | 13 | 13
score on a scale | 7.6 (1.5) | 7.0 (2.0)

4. Secondary Outcome: Heart Beat Abnormalities During Bowel Care (Number of Participants With Heart Beat Abnormalities)
Description: 3-lead electrocardiogram will be recorded throughout the duration of bowel care on two occasions within 28 days, for up to one hour on each occasion.
Time Frame: Measured continuously during bowel care (approximately one hour) on two occasions within 28 days.
Population: Proportion of participants reporting symptoms of palpitations during bowel care on each test day.
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Lubricant | Placebo Lubricant
Number analyzed (Participants) | 11 | 11
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: During the intervention (the duration of the bowel care program on each test day). Tests were conducted on 2 separate days within a 28 day period.
Groups:
- Lidocaine Lubricant Then Placebo Lubricant: In this arm, subjects will use lidocaine lubricant in their normal bowel care routine on day one and placebo lubricant on day two.
  Lidocaine lubricant: Subjects using this intervention will receive 30 mL of Lidocaine hydrochloride jelly (2%)
  Placebo lubricant: Subjects using this intervention will receive 30 mL of placebo lubricant (no topical anesthetic)
- Placebo Lubricant Then Lidocaine Lubricant.: In this arm, subjects will use regular lubricant (AMG MedPro lubricating gel) in their normal bowel care routine on day one and lidocaine lubricant on day two.
  Placebo lubricant: Subjects using this intervention will receive 30 mL of placebo lubricant (no topical anesthetic)
  Lidocaine lubricant: Subjects using this intervention will receive 30 mL of Lidocaine hydrochloride jelly (2%)
Arm/Group | Lidocaine Lubricant Then Placebo Lubricant | Placebo Lubricant Then Lidocaine Lubricant.
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT01567605/Prot_SAP_000.pdf